CLINICAL TRIAL: NCT07077863
Title: Transversus Abdominis Plane Block Applied by the Surgeon or Anaesthetist for Postoperative Pain Management in Gynaecological Cancer Surgery: a Retrospective Review
Brief Title: Transversus Abdominis Plane Block for Postoperative Pain Management in Gynaecological Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Duygu Akyol (Other Government)
Responsible Party: Sponsor-Investigator, Duygu Akyol, Principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Organization: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Other Study IDs: 2025-58
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Blocs
Keywords: gynecological cancer surgery; postoperative analgesia; transversus abdominis plane block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing gynecologic cancer surgery: Patients undergoing transversus abominis plan block for postoperative analgesia

SUMMARY:
The aim of this study was to compare the efficacy of transversus abdominis plane block for postoperative analgesia in gynaecological cancer surgery.

The main question(s) aimed to be answered are:

[For postoperative analgesia, a block performed by the surgeon in the area seen or a block performed by the anaesthetist before surgery?] Patients undergoing gynaecological cancer surgery were retrospectively reviewed. The investigators evaluated the effect of a four-quadrant transversus abdominis plane block for postoperative analgesia on pain scores and postoperative opioid use.

DETAILED DESCRIPTION:
This study was designed retrospectively. The investigators evaluated analgesia methods in patients undergoing surgery for gynaecological cancer between January 2024 and December 2024. The investigators evaluated the effect of transversus abdominis plane block on postoperative analgesia and opioid use.

ELIGIBILITY:
Inclusion Criteria:

* - Women aged 18 and over
* Gynaecological cancer surgery

Exclusion Criteria:

* - Patients undergoing peripheral or central block in addition to transversus abdominis plane block
* Allergy or history of local anaesthetic drug allergy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who underwent surgery for gynaecological cancer between January 2024 and December 2024 and to whom we applied four quadrant transversus abdominis plane block (TAPB) from peripheral nerve blocks for postoperative analgesia were included in the stud
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-07-12 (Actual)

PRIMARY OUTCOMES:
postoperative numerical rating scale | 24 hours postoperatively
  Our primary aim was to evaluate numerical rating scale at 24 hours postoperatively. numerical rating scale(NRS) was used to assess postoperative pain. NRS values were recorded For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: DUYGU AKYOL, M.D, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Basaksehir Cam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Ismail S, Siddiqui AS, Rehman A. Postoperative pain management practices and their effectiveness after major gynecological surgery: An observational study in a tertiary care hospital. J Anaesthesiol Clin Pharmacol. 2018 Oct-Dec;34(4):478-484. doi: 10.4103/joacp.JOACP_387_17. PMID 30774227
- [Background] Jakobsson J, Wickerts L, Forsberg S, Ledin G. Transversus abdominal plane (TAP) block for postoperative pain management: a review. F1000Res. 2015 Nov 26;4:F1000 Faculty Rev-1359. doi: 10.12688/f1000research.7015.1. eCollection 2015. PMID 26918134
- [Background] Bernard L, Lavecchia M, Trepanier G, Mah S, Pokoradi A, McGinnis JM, Alyafi M, Glezerson B, Nguyen J, Carlson V, Helpman L, Elit L, Jimenez W, Eiriksson L, Reade CJ. A double-blinded, randomized trial comparing surgeon-administered transversus abdominis plane block with placebo after midline laparotomy in gynecologic oncology surgery. Am J Obstet Gynecol. 2023 May;228(5):553.e1-553.e8. doi: 10.1016/j.ajog.2023.02.010. Epub 2023 Feb 14. PMID 36791986